CLINICAL TRIAL: NCT05243355
Title: A Prospective, Single-arm, Phase II Study of Envafolimab Combined With Chemotherapy and Recombinant Human Endostatin in the First-line Treatment of Advanced (Stage IIIB-IV) Squamous Non-small Cell Lung Cancer
Brief Title: Envafolimab Combined With Chemotherapy and Recombinant Human Endostatin in the First-line Treatment of Sq-NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMA-NSCLC-005
Record Dates: First submitted 2021-12-16; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2021-12

CONDITIONS: Squamous Non-small Cell Lung Cancer
MeSH Terms: interventions — envafolimab; Drug Therapy; Endostatins

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- "Envafolimab" and "Chemotherapy" and "Recombinant Human Endostatin" (Experimental): Envafolimab: 300 mg，D1，Q3W, until PD or intolerable toxicity. Paclitaxel / NAB-Paclitaxel, 175 / 260mg / m2, D1, Q3w. Cisplatin: 75mg / m2, 1-3 days, or carboplatin: AUC 5, D1, Q3w, 4-6 cycles. Recombinant Human Endostatin：210mg，CIV 72h，d1-3，Q3W，4-6 cycles in total.
  Interventions: Drug: "Envafolimab" and "Chemotherapy" and "Recombinant Human Endostatin"

INTERVENTIONS:
Drug: "Envafolimab" and "Chemotherapy" and "Recombinant Human Endostatin" — Envafolimab: 300 mg，D1，Q3W,until PD or intolerable toxicity Chemotherapy: Paclitaxel / NAB-Paclitaxel, 175 / 260mg / m2, D1, Q3w; Cisplatin: 75mg / m2, 1-3 days, or carboplatin: AUC 5, D1, Q3w, 4-6 cycles in total.
  Recombinant Human Endostatin：210mg，CIV 72h，d1-3，Q3W，4-6 cycles in total.

SUMMARY:
This is a prospective, single arm, multicenter phase II study aimed at evaluating the efficacy and safety of Envafolimab combined with standard platinum containing dual drug chemotherapy and Recombinant Human Endostatin in patients with advanced (stage IIIB-IV) squamous non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent；
* Aged 18-75 years old；
* Histologically or cytologically confirmed, locally advanced (Stage IIIB/C) not amenable to curative surgery or radiotherapy, or metastatic/recurrent (Stage IV) squamous NSCLC according to American Joint Committee on Cancer, 8th Edition；
* At least 1 measurable lesion as defined by RECIST v1.1；
* ECOG performance status 0-1；
* No systematic antitumor treatment for advanced / metastatic diseases has been received in the past；
* Life expectancy sup 3 months；
* Adequate organ function；
* For female subjects of childbearing age, urine or serum pregnancy test shall be conducted 3 days before receiving the first study drug administration, and the result is negative；
* The subject and the subject's sexual partner need to use a medically approved contraceptive measure during the study treatment period and within 6 months after the end of the study treatment period.

Exclusion Criteria:

* Histology was non squamous cell NSCLC. Mixed cell types must distinguish the dominant cell morphology (squamous cell carcinoma components > 50% can be included in the group); If there are small cell carcinoma, neuroendocrine carcinoma and sarcoma, they can not be included in the group;
* EGFR sensitive mutations or ALK rearrangements;
* Imaging (CT or MRI) showed that the tumor invaded large blood vessels or it was judged that the tumor was very likely to invade important blood vessels and cause fatal bleeding during the follow-up study;
* Concurrent participation in another clinical trial;
* Have previously received the following therapies: anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or drugs that stimulate or co inhibit T cell receptors (e.g., CTLA-4, OX-40, CD137);
* Received Chinese patent medicine with anti-tumor indications or drugs with immunomodulatory effect (thymosin, interferon, interleukin, etc.) within 2 weeks, or major surgical treatment within 3 weeks before the first administration;
* There are active hemoptysis, active diverticulitis, abdominal abscess, gastrointestinal obstruction and peritoneal metastasis that need clinical intervention;
* Grade III-IV congestive heart failure (New York Heart Association classification), poorly controlled and clinically significant arrhythmia;
* Any arterial thrombosis, embolism or ischemia, such as myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack, occurred within 6 months before enrollment;
* Known allergic reactions to PD-1/L1 monoclonal antibodies, taxanes, cisplatin or carboplatin, recombinant human endostatin active ingredients and or any excipients;
* Patients requiring long-term systemic use of corticosteroids;
* Symptomatic central nervous metastasis;
* Active infection requiring treatment or systemic anti infective drugs used within one week before the first administration;
* Not fully recovered from toxicity and/or complications caused by any intervention before starting treatment (i.e. ≤ grade 1 or reaching baseline, excluding fatigue or hair loss);
* Known HIV infection;
* Untreated active hepatitis B (defined as HBsAg positive and HBV-DNA copy number detected greaterthan the upper limit of normal value in the laboratory of the research center);
* Active HCV infected;
* Live vaccine was administered within 30 days before the first administration;
* Pregnant or lactating women;
* Medical history or disease evidence, abnormal treatment or laboratory test values that may interfere with the test results, prevent the subjects from participating in the whole study, or other situations that the researchers believe are not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-12-03 (Actual); Primary Completion 2023-12-03 (Estimated); Study Completion 2024-12-03 (Estimated)

PRIMARY OUTCOMES:
1 year PFS rate | 12 months after the last subject participating in
  12-month progression free survival in ITT population

SECONDARY OUTCOMES:
ORR | 24 months after the last subject participating in
  The proportion of subjects with complete response (CR) and partial response (PR) in total subjects
DOR | 24 months after the last subject participating in
  DoR (per RECIST 1.1) is defined as the time from the date for first documented response of complete response (CR) or partial response (PR) to the date of first documented of disease progression or death, whichever occurs first.
PFS | 24 months after the last subject participating in
  Progression-free survival (PFS per RECIST 1.1) is defined as the time from the starting date of study drug to the date of first documentation of disease progression or death, whichever occurs first
OS | 24 months after the last subject participating in
  OS is defined as the time from the starting date of study drug to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Qilu hospital of Shandong univertisy, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan

IPD SHARING:
Plan to Share IPD: No